CLINICAL TRIAL: NCT02689440
Title: Therapy of Early Chronic Phase Chronic Myelogenous Leukemia (CML) With Dasatinib and Venetoclax: A Phase II Study
Brief Title: Dasatinib and Venetoclax in Treating Patients With Philadelphia Chromosome Positive or BCR-ABL1 Positive Early Chronic Phase Chronic Myelogenous Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1040; NCI-2016-00362 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-1040 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Philadelphia Chromosome Positive, BCR-ABL1 Positive Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dasatinib, venetoclax) (Experimental): Patients receive dasatinib PO QD for 15 years in the absence of disease progression or unacceptable toxicity. After 3 months of dasatinib treatment, patients also receive venetoclax PO QD on days 1-14 of each month for 3 years in the absence of disease progression or unacceptable toxicity (patients enrolled prior to 4/1/2018 receive only dasatinib).
  Interventions: Drug: Dasatinib; Other: Laboratory Biomarker Analysis; Drug: Venetoclax

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well dasatinib and venetoclax work in treating patients with Philadelphia chromosome positive or BCR-ABL1 positive early chronic phase chronic myelogenous leukemia. Dasatinib and venetoclax may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients with previously-untreated chronic phase chronic myeloid leukemia (CML) who achieve major molecular response by 12 months of treatment with dasatinib 50 mg orally daily (first 70 patients) and of dasatinib 50 mg daily in combination with venetoclax 200 mg daily starting after 3 months of dasatinib therapy (after protocol amendment).

SECONDARY OBJECTIVES:

I. To estimate the 12 months molecular response (MR)4.5 rate and the cumulative overall rate of MR4.5 (BCR-ABL transcripts [IS] =< 0.01%).

II. To estimate the proportion of patients with MR4.5 at 6-, 12-, 18-, 24-, and 36-months of therapy.

III. To estimate the proportion of patients with sustained MR4.5 of 3 years and more.

IV. To estimate the treatment-free remission rate, time to progression, and overall survival.

V. To assess the safety of this combination.

OUTLINE:

Patients receive dasatinib orally (PO) once daily (QD) for 15 years in the absence of disease progression or unacceptable toxicity. After 3 months of dasatinib treatment, patients also receive venetoclax PO QD on days 1-14 of each month for 3 years in the absence of disease progression or unacceptable toxicity (patients enrolled prior to 4/1/2018 receive only dasatinib).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ph-positive or BCR-ABL positive CML in early chronic phase CML (i.e., time from diagnosis ≤ 12 months). Except for hydroxyurea and/or 1 to 2 doses of cytarabine patients must have received no or minimal prior therapy, defined as <1 month (30 days) of prior FDA approved TKI.

  * Clonal evolution defined as the presence of additional chromosomal abnormalities other than the Ph chromosome has historically been included as a criterion for accelerated phase. However, patients with clonal evolution as the only criterion of accelerated phase have a significantly better prognosis, and when present at diagnosis may not impact the prognosis at all. Thus, patients with clonal evolution and no other criteria for accelerated phase will be eligible for this study.
* Eastern Cooperative Oncology Group (ECOG) performance of 0-2
* Total bilirubin < 1.5 x upper limit normal (ULN) (unless secondary to Gilbert's disease, in which case should be < 2.5x ULN)
* Serum glutamate pyruvate transaminase (SGPT) < 3 x ULN
* Creatinine < 1.5 x ULN
* Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital

Exclusion Criteria:

* New York Heart Association (NYHA) cardiac class 3-4 heart disease
* Patients meeting the following criteria are not eligible unless cleared by cardiology:

  * Uncontrolled angina within 3 months
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  * Prolonged QTc interval on pre-entry electrocardiogram (> 460 msec)
  * History of significant bleeding disorder unrelated to cancer, including:

    * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
    * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Patients with active, uncontrolled psychiatric disorders include: psychosis, major depression, and bipolar disorders
* Subject is known to be positive for human immunodeficiency virus (HIV); (HIV testing is not required)
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
  * Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
* Women of pregnancy potential must practice an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Women must continue birth control for the duration of the trial and at least 3 months after the last dose of study drug.

Pregnant or breast-feeding women are excluded. All WOCBP must have a negative pregnancy test prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive study drug and must not be enrolled in the study.

* Patients in late chronic phase (i.e., time from diagnosis to treatment > 12 months), accelerated or blast phase are excluded; the definitions of CML phases are as follows:

  * Early chronic phase:

    * Time from diagnosis to therapy ≤12 months
    * Late chronic phase:

      * Time from diagnosis to therapy > 12 months
  * Blastic phase:

    * Presence of 30% blasts or more in the peripheral blood or bone marrow
  * Accelerated phase CML:

    * Presence of any of the following features:

      * Peripheral or marrow blasts 15% or more
      * Peripheral or marrow basophils 20% or more
      * Thrombocytopenia < 100 x 10^9/L unrelated to therapy
      * Documented extramedullary blastic disease outside liver or spleen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Major molecular response (MMR) defined as BCR-ABL transcripts (IS) =< 0.1% | Up to 12 months
  MMR estimates will be presented with 95% credible intervals. MMR and patient and clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test.

SECONDARY OUTCOMES:
Complete cytogenetic response (CCR) defined as 0% Ph-positive metaphases, or fluorescence in situ hybridization =< 2%, or BCR-ABL transcripts (IS) =< 1% | At 6 months
  CCR estimates will be presented with 95% credible intervals.
Incidence of toxicities, defined as grade 3 or higher pleural effusion | Up to 3 years
  Safety data of the patients will be summarized using descriptive statistics such as mean, standard deviation, median and range (i.e., duration of hematologic, cytogenetic and molecular response to the drug).
Time to progression | Up to 3 years
  Estimated using the Kaplan-Meier method. The two-sided log-rank test will be used to assess the differences of time to events between groups.
Overall survival | Up to 3 years
  Estimated using the Kaplan-Meier method. The two-sided log-rank test will be used to assess the differences of time to events between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gener-Ricos G, Haddad FG, Sasaki K, Issa GC, Skinner J, Masarova L, Borthakur G, Alvarado Y, Garcia-Manero G, Jabbour E, Kantarjian H. Low-Dose Dasatinib (50 mg Daily) Frontline Therapy in Newly Diagnosed Chronic Phase Chronic Myeloid Leukemia: 5-Year Follow-Up Results. Clin Lymphoma Myeloma Leuk. 2023 Oct;23(10):742-748. doi: 10.1016/j.clml.2023.05.009. Epub 2023 May 23. PMID 37308342
- [Derived] Naqvi K, Jabbour E, Skinner J, Anderson K, Dellasala S, Yilmaz M, Ferrajoli A, Bose P, Thompson P, Alvarado Y, Jain N, Takahashi K, Burger J, Estrov Z, Borthakur G, Pemmaraju N, Paul S, Cortes J, Kantarjian HM. Long-term follow-up of lower dose dasatinib (50 mg daily) as frontline therapy in newly diagnosed chronic-phase chronic myeloid leukemia. Cancer. 2020 Jan 1;126(1):67-75. doi: 10.1002/cncr.32504. Epub 2019 Sep 25. PMID 31553487
- [Derived] Naqvi K, Jabbour E, Skinner J, Yilmaz M, Ferrajoli A, Bose P, Thompson P, Alvarado Y, Jain N, Takahashi K, Burger J, Estrov Z, Borthakur G, Pemmaraju N, Paul S, Cortes J, Kantarjian HM. Early results of lower dose dasatinib (50 mg daily) as frontline therapy for newly diagnosed chronic-phase chronic myeloid leukemia. Cancer. 2018 Jul 1;124(13):2740-2747. doi: 10.1002/cncr.31357. Epub 2018 May 3. PMID 29723397
- See also: MD Anderson Cancer Center — http://www.mdanderson.org